CLINICAL TRIAL: NCT03641508
Title: Long Term Effectiveness of Trigger Finger Injections With Triamcinolone vs. Dexamethasone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ericka Lawler (Other)
Responsible Party: Sponsor-Investigator, Ericka Lawler, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201308766
Record Dates: First submitted 2017-08-04; First posted 2018-08-22 (Actual); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Trigger Finger Disorder
Keywords: trigger finger
MeSH Terms: conditions — Trigger Finger Disorder | interventions — Triamcinolone; Triamcinolone Acetonide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triamcinolone (Active Comparator): The study drug used will be triamcinolone mixed with 1% lidocaine without epinephrine
  Interventions: Drug: Triamcinolone
- Dexamethasone (Active Comparator): The study drug used will be dexamethasone mixed with 1% lidocaine without epinephrine
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Triamcinolone — Triamcinolone acetonide (Kenalog; 10 mg/mL; insoluble). This will be mixed with 1% lidocaine without epinephrine
  Other Names: Kenalog
  Arms: Triamcinolone
Drug: Dexamethasone — dexamethasone sodium phosphate (Decadron; 4 mg/mL; soluble). Again, this will be mixed with 1% lidocaine without epinephrine
  Other Names: Decadron
  Arms: Dexamethasone

SUMMARY:
Trigger finger (stenosing tenosynovitis) is a very common condition and in office treatment with corticosteroid injection is widely accepted to be first line treatment. Previous studies have reported resolution of triggering after injection at rates ranging from 50% to 93%. Many factors contribute to this variability, including duration of symptoms, presence of diabetes, etc. This study will be a single center, prospective, randomized control trial. Patients will be collected into two different cohorts. The main cohort will be of patients with primary, idiopathic trigger finger. A second cohort of patients with diabetes will also be collected for secondary study questions. Study procedures will include clinical examination of the patient, injection of trigger fingers with mix of local anesthetic and one of two steroids, possible repeat trigger finger injections, and if patients are so indicated, surgical treatment of the trigger finger. Surgical treatment is considered clinical care of these patients who have continued or recurrent symptoms and the surgical treatment would not be considered part of this study. During the study, patients will also fill out surveys about their symptoms. The study drugs used will be 1% lidocaine without epinephrine mixed with either triamcinolone or dexamethasone. These medications are FDA approved for injection treatment of "acute non-specific tenosynovitis." This indication includes trigger finger which is also known as acute stenosing tenosynovitis. The package inserts listing the indications for use of these medications are included in the attachments portion of the IRB application.

DETAILED DESCRIPTION:
Upon coming to a clinical visit, patients who are complaining of trigger finger will be asked if they would like to participate in a study. After finishing the consent process, patients who elect to participate will be randomized to one of the two steroid groups. All patients will complete an initial enrollment survey as well as a DASH score (Disabilities of the Arm, Shoulder, and Hand), and the Michigan Hand Questionnaire (MHQ). Each patient will be examined by one of the attending physicians or one of the experienced physician's assistants and their Quinnell grade of trigger finger will be documented. Injection will performed in a standardized fashion in clinic. Multiple trigger fingers in any one patient will be treated but patients will be randomized, not individual fingers. The most radial finger treated will be the one followed for outcome measures. Patients will have the option to be treated with a different medication if they require further injections. However, all patients and data will be analyzed in an intention to treat manner. Follow-up visits will be arranged at 6 weeks, 6 months, 1 year, and 2 years. At each follow-up visit, patients will again fill out the DASH score, MHQ, and a study-specific survey to evaluate outcome. In anticipation of the difficulty of obtaining a high follow-up rate at the 1 year and 2 year marks, the study-specific survey and the DASH and the MHQ may be administered to the patients over the phone or be sent an electronic version of the surveys. Additionally, these patients will also receive a written copy of the surveys via mail to complete and return. All patients will be followed for a total of 2 years after their latest injection. Most of these procedures are standard of care, the only research visits are the 1 and 2 year follow-up visits. Some patients with recurrent or continued symptoms may be indicated for surgical treatment of their trigger finger. Surgical treatment is considered clinical care of these patients who have continued or recurrent symptoms and the surgical treatment would not be considered part of this study.

Data collected from the patient's medical record will include demographic information such as age, sex, birthdate. The investigators will also review whether the patient is currently taking any medications for the treatment of diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed primary, idiopathic trigger finger(s)
* Quinnell grade II or greater.
* Patients must be 18 years of age or older

Exclusion Criteria:

* patients taking any diabetic medications.
* any history of inflammatory or autoimmune arthritis
* history of prior trauma to the tendon of the affected digit
* pregnancy, and breast feeding

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ericka Lawler, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freiberg A, Mulholland RS, Levine R. Nonoperative treatment of trigger fingers and thumbs. J Hand Surg Am. 1989 May;14(3):553-8. doi: 10.1016/s0363-5023(89)80024-3. PMID 2738345
- [Background] Griggs SM, Weiss AP, Lane LB, Schwenker C, Akelman E, Sachar K. Treatment of trigger finger in patients with diabetes mellitus. J Hand Surg Am. 1995 Sep;20(5):787-9. doi: 10.1016/S0363-5023(05)80432-0. PMID 8522745
- [Background] Lapidus PW, Guidotti FP. Stenosing tenovaginitis of the wrist and fingers. Clin Orthop Relat Res. 1972 Mar-Apr;83:87-90. doi: 10.1097/00003086-197203000-00015. No abstract available. PMID 5014835
- [Background] Marks MR, Gunther SF. Efficacy of cortisone injection in treatment of trigger fingers and thumbs. J Hand Surg Am. 1989 Jul;14(4):722-7. doi: 10.1016/0363-5023(89)90199-8. PMID 2754207
- [Background] Murphy D, Failla JM, Koniuch MP. Steroid versus placebo injection for trigger finger. J Hand Surg Am. 1995 Jul;20(4):628-31. doi: 10.1016/S0363-5023(05)80280-1. PMID 7594291
- [Background] Newport ML, Lane LB, Stuchin SA. Treatment of trigger finger by steroid injection. J Hand Surg Am. 1990 Sep;15(5):748-50. doi: 10.1016/0363-5023(90)90149-l. PMID 2229972
- [Background] Rhoades CE, Gelberman RH, Manjarris JF. Stenosing tenosynovitis of the fingers and thumb. Results of a prospective trial of steroid injection and splinting. Clin Orthop Relat Res. 1984 Nov;(190):236-8. PMID 6488636
- [Background] Ring D, Lozano-Calderon S, Shin R, Bastian P, Mudgal C, Jupiter J. A prospective randomized controlled trial of injection of dexamethasone versus triamcinolone for idiopathic trigger finger. J Hand Surg Am. 2008 Apr;33(4):516-22; discussion 523-4. doi: 10.1016/j.jhsa.2008.01.001. PMID 18406955
- [Background] Stahl S, Kanter Y, Karnielli E. Outcome of trigger finger treatment in diabetes. J Diabetes Complications. 1997 Sep-Oct;11(5):287-90. doi: 10.1016/s1056-8727(96)00076-1. PMID 9334911
- [Background] Wolfe, Scott W. "Chapter 62-Tendinopathy." Green's Operative Hand Surgery, 6th Ed. Elsevier, Philadelphia. 2011.

RESULTS

PARTICIPANT FLOW:
Period: First Injection
Arm/Group | Triamcinolone | Dexamethasone
Started | 37 | 32
Completed | 35 | 32
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: Follow-up/Second Injection
Arm/Group | Triamcinolone | Dexamethasone
Started (Only those who had symptoms at the six-week follow-up received the second injection) | 2 | 10 (Only those who had symptoms at the six-week follow-up received the second injection)
Completed | 2 (Only those who had symptoms at the six-week follow-up received the second injection) | 10 (Only those who had symptoms at the six-week follow-up received the second injection)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triamcinolone | Dexamethasone | Total
Number analyzed (Participants) | 37 | 32 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (8.55) | 63.7 (11.37) | 61.94 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 10 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 37 | 32 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Symptoms of Trigger Finger
Description: Number of participants with no symptoms of trigger finger 6 weeks after the initial encounter for both groups. Outcomes were determined clinically:
  The Quinnell grading system was used for objectively evaluating the trigger finger. This grading system is a scale of 0-4 for severity of triggering with 0 being no triggering.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone | Dexamethasone
Number analyzed (Participants) | 35 | 32
Participants | 28 | 9

2. Primary Outcome: Number of Participants With no Symptoms of Trigger Finger
Description: Number of participants with no symptoms of trigger finger 6 months after the initial encounter for both groups. Outcomes were determined clinically:
  The Quinnell grading system was used for objectively evaluating the trigger finger. This grading system is a scale of 0-4 for severity of triggering with 0 being no triggering.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone | Dexamethasone
Number analyzed (Participants) | 35 | 32
Participants | 23 | 12

3. Primary Outcome: Number of Participants With no Symptoms of Trigger Finger
Description: Number of participants with no symptoms of trigger finger 1 year after the initial encounter for both groups. Outcomes were determined clinically:
  The Quinnell grading system was used for objectively evaluating the trigger finger. This grading system is a scale of 0-4 for severity of triggering with 0 being no triggering.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Triamcinolone | Dexamethasone
Number analyzed (Participants) | 35 | 32
Participants | 20 | 13

ADVERSE EVENTS:
Arm/Group | Triamcinolone | Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/32
Other Adverse Events (participants affected / at risk) | 10/37 | 7/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone (N=37) | Dexamethasone (N=32)
Transient numbness (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5)
Pigment change (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes